CLINICAL TRIAL: NCT05686408
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy, Safety, and Tolerability of TNX-601 ER Monotherapy Versus Placebo in Patients With Major Depressive Disorder (MDD)
Brief Title: Study to Evaluate TNX-601 ER Monotherapy Versus Placebo in Patients With Major Depressive Disorder (MDD)
Acronym: UPLIFT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Collaborators: Rho, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNX-TI-M201
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Depression; Depressive Disorder; Depressive Symptoms; Depressive Disorder, Major; Depressive Episode; Depression Severe
MeSH Terms: conditions — Depression; Depressive Disorder; Depressive Disorder, Major | interventions — tianeptine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TNX-601 ER, 39.4 mg (Experimental): 1x TNX-601 ER, 39.4 mg, tablet taken orally once daily for 6 weeks.
  Interventions: Drug: TNX-601 ER
- Placebo (Placebo Comparator): Placebo tablet taken orally once daily for 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TNX-601 ER — Patients will take 1 tablet orally once daily for 6 weeks.
  Other Names: Tianeptine
  Arms: TNX-601 ER, 39.4 mg
Drug: Placebo — Patients will take 1 tablet orally once daily for 6 weeks.
  Arms: Placebo

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy, safety, and tolerability of TNX-601 ER monotherapy versus placebo in patients with Major Depressive Disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* Female or male aged 18 to 65 years (inclusive).
* Have a primary DSM-5 diagnosis of current MDD.

  1. The duration of the current MDE must be at least 12 weeks.
  2. Without psychotic or catatonic features.

Exclusion Criteria:

* Psychiatric History:

  1. Diagnosis of DSM-5-defined lifetime bipolar disorder (I, II, or unspecified), schizophrenia, schizoaffective disorder, MDD with psychotic features, other psychotic disorder, or antisocial personality disorder; current (past month) obsessive-compulsive disorder; current (past month) posttraumatic stress disorder; current (past 3 months) anorexia nervosa; lifetime opioid or lifetime sedative-hypnotic use disorders, as confirmed by the MINI 7.0.2.
  2. Diagnosis of borderline personality disorder
  3. Patients with comorbid generalized anxiety disorder (GAD), social anxiety disorder (SAD), or panic disorder are excluded only if the GAD, SAD, or panic disorder is considered the primary psychiatric diagnosis, rather than MDD. (If MDD is the primary diagnosis, patients with comorbid GAD, SAD, and panic disorder are allowed for randomization).
* Patients with treatment refractory MDD, ie, previously having in their lifetime failed ≥2 treatments with at least 2 different classes of antidepressants of adequate dose, duration, and treatment adherence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Sullivan, MD, Study Director — Tonix Pharmaceuticals
Locations (27):
- United States (27):
  - Preferred Research Partners, Little Rock, Arkansas
  - Cenexel CIT - Bellflower, Bellflower, California
  - Behavioral Research Specialists, Glendale, California
  - Synergy Research, Lemon Grove, California
  - Excell Research, Oceanside, California
  - NCR Research Institute, Orange, California
  - Cenexel CIT - Riverside, Riverside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Cenexel CNR - Sherman Oaks, Sherman Oaks, California
  - Viking Clinical Research, Temecula, California
  - Mountain View Clinical Research, Denver, Colorado
  - CT Clinical Research Associates, Cromwell, Connecticut
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Clinical Neuroscience Solutions - Jacksonville, Jacksonville, Florida
  - West Broward Outpatient Clinic, Lauderhill, Florida
  - Segal Trials - North Miami, Miami Lakes, Florida
  - Clinical Neuroscience Solutions - Orlando, Orlando, Florida
  - Cenexel ACMR - Atlanta, Atlanta, Georgia
  - Cenexel Research - Decatur, Decatur, Georgia
  - Northwest Clinical Trials, Boise, Idaho
  - Chicago Research Center, Chicago, Illinois
  - Cenexel HRI - Berlin, Berlin, New Jersey
  - Summit Research Network, Portland, Oregon
  - Clinical Neuroscience Solutions - Memphis, Memphis, Tennessee
  - Donald J. Garcia, Jr., Austin, Texas
  - Futuresearch Trials of Dallas, Dallas, Texas
  - Core Clinical Research, Everett, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | TNX-601 ER, 39.4 mg
Started | 68 | 64
Completed | 58 | 53
Not Completed | 10 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TNX-601 ER, 39.4 mg | Total
Number analyzed (Participants) | 68 | 64 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (13.87) | 40.2 (11.92) | 41.0 (12.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 38 | 77
  Male | 29 | 26 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 16 | 28
  Not Hispanic or Latino | 56 | 48 | 104
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 14 | 33
  White | 44 | 45 | 89
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 68 | 64 | 132

OUTCOME MEASURES:

1. Primary Outcome: Montgomery Asberg Depression Rating Scale (MADRS)
Description: Change from Baseline (Visit 2) in the MADRS total score at Week 6. Scores range from 0 to 60. Lower scores indicate less depression.
Time Frame: Day 1 and Week 6
Population: Results reported for ITT population, which includes all randomized patients who received at least one dose of IP.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TNX-601 ER, 39.4 mg
Number analyzed (Participants) | 68 | 64
units on a scale | -12.8 (1.32) | -12.7 (1.30)

2. Secondary Outcome: Clinical Global Impression of Severity (CGI-S)
Description: Change from Baseline (Visit 2) in the Clinical Global Impression of Severity Scale (CGI-S) score at Week 6. Scores range from 1 to 7. Lower scores indicate less severe illness.
Time Frame: Day 1 and Week 6
Population: Results reported for ITT population, which includes all randomized patients who received at least one dose of IP.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TNX-601 ER, 39.4 mg
Number analyzed (Participants) | 68 | 64
units on a scale | -1.2 (0.16) | -1.0 (0.15)

3. Secondary Outcome: Sheehan Disability Scale (SDS)
Description: Change from Baseline (Visit 2) in the Sheehan Disability Scale (SDS) total score at Week 6. Scores range from 0 to 30. Lower scores indicate less impairment to activities.
Time Frame: Day 1 and Week 6
Population: Results reported for ITT population, which includes all randomized patients who received at least one dose of IP.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TNX-601 ER, 39.4 mg
Number analyzed (Participants) | 68 | 64
units on a scale | -7.3 (0.97) | -5.8 (0.95)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Placebo | TNX-601 ER, 39.4 mg
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/64
Serious Adverse Events (participants affected / at risk) | 1/68 | 2/64
Other Adverse Events (participants affected / at risk) | 3/68 | 7/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=68) | TNX-601 ER, 39.4 mg (N=64)
Seizure (Nervous system disorders) | 0 | 1
Generalized tonic-clonic seizure (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=68) | TNX-601 ER, 39.4 mg (N=64)
Nausea (Gastrointestinal disorders) | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An industry standard NDA is in place with all investigators.

DOCUMENTS (2):
  • Study Protocol (2023-03-02): https://cdn.clinicaltrials.gov/large-docs/08/NCT05686408/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/08/NCT05686408/SAP_001.pdf